CLINICAL TRIAL: NCT05947344
Title: A Multicenter, Open, Dose Escalation and Dose Expansion Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of STI-8591 in Subjects With Advanced Acute Myeloid Leukemia (AML)
Brief Title: A Study to Evaluate the STI-8591 in Subjects With Advanced Acute Myeloid Leukemia (AML)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLT3-AML-101CN
Record Dates: First submitted 2023-06-25; First posted 2023-07-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: AML, Adult
Keywords: FLT3 inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- STI-8591 in Advanced Acute Myeloid Leukemia (AML) (Experimental): Subjects with Advanced primary AML or MDS secondary to AML or AML-MR.
  Interventions: Drug: STI-8591

INTERVENTIONS:
Drug: STI-8591 — Four dosing cohorts will be evaluated in the dose escalation phase: 20mg, 40mg, 60mg and 80mg. Expansion is planned in two dose groups of 40mg and 60mg.
  Other Names: STI-8591 alone

SUMMARY:
This is a first-in-human, dose-escalation and dose-expansion Phase I study to evaluate the safety, tolerability, pharmacokinetics (PK) and efficacy of STI-8591 in subjects with advanced AML who have signed an informed consent form (ICF) and have been screened for enrollment in this study.

* Dose escalation phase: rapid titration and conventional 3+3 test design were used to evaluate the safety, dose-limiting toxicity (DLT), maximum tolerated dose (MTD) and PK characteristics of STI-8591.
* Dose Expansion Phase: Evaluate the safety, preliminary efficacy and determine the recommended phase II dose (RP2D) of STI-8591 for the treatment of subjects with advanced AML under the conditions of reaching the expanded dose.

DETAILED DESCRIPTION:
Dose escalation phase:Based on the preclinical trial data and with reference to the modified Fibonacci method, the dose escalation ratios are 100%, 100%, 50% and 6.7%, and the initial 5 dose groups for STI-8591 dose escalation are 40, 80, 160, 240 and 280 mg/day, respectively. Screened subjects will be entered into the 5 dose groups in order of succession from lowest to highest dose.This test dose increment will be performed using the rapid titration method and the traditional 3+3 test design.

Dose expansion phase:During dose escalation, for dose groups (except for ≥2 DLT dose groups) when the following dose signals suggesting initial efficacy are present.

1) CR, CRh or CRi in ≥1 subject in either dose group.2) Median decrease in FLT3 phosphorylation was ≥90% in ≥3 subjects in either dose group.The SRC will decide whether to initiate an extension study for that dose group and its subsequent dose groups at the same time as the dose escalation to the next dose group. Subjects in the dose escalation phase will be administered BID every 28 days in 1 cycle, with ≥8h between doses, fasting for at least 2 hours before and at least 1 hour after dosing with approximately 240mL of water (subject to adjustment based on data results from the dose escalation phase) . If initiation was determined, the dose group identified for initiation and its subsequent dose group extension studies were further enrolled in 14 to 17 cases [a total of 20 cases in each dose group, with FLT3 mutation-positive (FLT3 internal tandem repeat (ITD) and/or FLT3 tyrosine kinase structural domain (TKD) mutation-positive subjects enrolled in at least 10 cases] to further define the final RP2D.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in this study, subjects must meet all of the following inclusion criteria.

1. Voluntary signing of ICF.
2. Age ≥ 18 years old.
3. Expected survival >12 weeks.
4. Dose escalation component: Advanced primary AML or myelodysplastic neoplasm (MDS) secondary to AML or MDS/myeloproliferative neoplasm (MPN)-associated AML (AML-MR) diagnosed by 2022 WHO AML typing and with diagnostic criteria that have failed standard therapy or are intolerant of standard therapy may be considered for inclusion in this component of the study. Dose extension section: Advanced primary AML or MDS secondary to AML or AML-MR diagnosed according to the 2022 WHO AML typing and associated diagnostic criteria, who have failed or are intolerant to standard therapy, or who are unable to access standard therapy for various reasons, may only be considered for inclusion in this part of the study.
5. ECOG scores physical fitness status 0 to 2.
6. Subjects are willing to undergo a bone marrow aspiration/biopsy as required by the protocol, which is used to assess the subject's response to treatment.
7. Laboratory test index requirements within 7 days prior to the first dose, including:

   White blood cell count (WBC) ≤ 20 x 109 /L [(hydroxyurea is allowed up to the first dose to stabilize the WBC count up to a maximum dose of 5 g/day. Hydroxyurea may be continued for up to 28 days after the first dose (i.e., the first dosing cycle) at the discretion of the investigator, but generally not beyond 28 days)].

   Alanine aminotransferase (ALT) ≤ 2.5 x ULN (≤ 5 x ULN if liver involvement is known).

   Aspartate aminotransferase (AST) ≤ 2.5 x ULN (≤ 5 x ULN if liver involvement is known) Total bilirubin (TBIL) ≤ 1.5 x ULN (< 3.0 x ULN if diagnosed with Gilbert's syndrome) Estimated glomerular filtration rate (eGFR, calculated according to the Cockcroft-Gault formula or by measuring 24-hour urine) > 50 mL/min.
8. Residual toxicity of previous antitumor therapy ≤ grade 1 (except alopecia and hyperpigmentation; see inclusion criteria 7 for laboratory test indices)
9. Be willing and able to comply with the study schedule and all other study protocol requirements.
10. Women of childbearing potential (WOCBP) (women of childless potential defined as sexually mature women who have undergone hysterectomy or bilateral oophorectomy or bilateral salpingo-oophorectomy or bilateral tubal ligation/closure, or who are unable to have children because of congenital or acquired disease or who have been spontaneously menopausal for ≥12 months) must have a negative blood pregnancy test performed during screening.
11. Female subjects of childbearing potential and male subjects whose partners are of childbearing potential must use a highly effective method of contraception from the time of screening until 180 days after the last treatment.
12. Subjects are required to provide FLT3 mutation status testing within 6 months prior to the first dose, and if not, are willing to undergo screening period testing as required by the protocol.

Exclusion Criteria:

To be enrolled in this study, subjects must not meet any of the following exclusion criteria.

1. Known hypersensitivity to any component of the study drug formulation.
2. Subjects were diagnosed with acute promyelocytic leukemia (APL).
3. Subjects have BCR-ABL positive leukemia (chronic myelogenous leukemia acute).
4. Subjects developed secondary AML after previous antitumor therapy for other tumors (except MDS, MDS/MPN).
5. Subjects had CNS leukemia with associated clinical symptoms.
6. Enrolled in any therapeutic clinical study within 28 days prior to the first dose and enrolled in treatment, except in the survival follow-up phase of the interventional study.
7. Received anti-tumor therapy (including chemotherapy, immunotherapy, endocrine therapy, targeted therapy, etc.) within 28 days or 5 half-lives (whichever is shorter) prior to the first dose. Received radiotherapy within 14 days prior to the first dose. Palliative radiotherapy for symptom control is allowed to be completed at least 7 days prior to the first dose. Have received herbal therapy with approved indications for antitumor use within 7 days prior to the first dose.
8. ≥ Grade 2 graft-versus-host disease (GvHD), including acute, chronic or overlapping or escalating GvHD therapy within 14 days prior to first dose or being treated with systemic cortisol hormone for GvHD.
9. Received chimeric antigen receptor T-cell immunotherapy (CAR-T) within 3 months prior to the first dose.
10. Strong inducer or strong inhibitor of cytochrome P450 (CYP450) 2C8 or 3A4 enzymes taken within 14 days prior to the first dose, unless the investigator assesses that the drug is necessary for the subject's treatment regimen.
11. Major surgery within 28 days prior to first dose or minor surgery within 7 days prior to first dose, except diagnostic biopsy, insertion of vascular access device
12. Subjects have clinically significant coagulation abnormalities, such as disseminated intravascular coagulation (DIC), hemophilia A, hemophilia B, and vascular hemophilia.
13. Intractable hypokalemia or hypomagnesemia that is not easily corrected by symptomatic treatment and with previous recurrent episodes.
14. Active tuberculosis, or interstitial lung disease requiring corticosteroid therapy, drug-induced interstitial lung disease, history of radiation pneumonia, or clinically active interstitial lung disease as suggested by any current evidence, prior to the first dose.
15. Presence of an uncontrolled active infection (defined as exhibiting persistent signs/symptoms associated with the infection that do not improve despite appropriate antibiotic or other treatment) within 72 hours prior to the first dose. Ongoing use of prophylactic antibiotics, antifungals, or antivirals is eligible for enrollment.
16. Inability to take oral medication, history of previous surgery or severe gastrointestinal disorders such as dysphagia and active gastric ulcer, which the investigator believes may affect the absorption of the study drug.
17. History of deep vein thrombosis, pulmonary embolism, or any other serious thromboembolism (other than thrombosis due to vascular access devices or superficial venous thrombosis) within 3 months prior to the first dose.
18. Active or uncontrolled HBV (HBsAg positive and/or HBcAb positive with positive HBV-DNA titers), HCV (HCV-Ab positive with positive HCV-RNA titers), HIV positive.
19. History of clinically significant cardiovascular disease, including.

    1. Congestive heart failure (NYHA classification ≥ Class III) within 6 months prior to first dose
    2. Unstable angina occurred within 6 months prior to the first dose.
    3. Myocardial infarction within 6 months prior to the first dose.
    4. Presence of poorly controlled arrhythmias at screening (e.g., subjects with ventricular tachycardia occurring during antiarrhythmic drug therapy will be excluded; however, subjects with atrioventricular block of degree I or asymptomatic left anterior bundle branch block/right bundle branch block do not have to be excluded).
    5. Diagnosis or suspicion of long QT syndrome at screening (including a family history of long QT syndrome)
    6. QTcF interval >450 msec (using the Fridericia formula).
    7. Left ventricular ejection fraction (LVEF) <45%.
    8. Uncontrolled hypertension (on the basis of lifestyle improvement, blood pressure has not reached the standard after applying a reasonably tolerable adequate dose of 2 or more antihypertensive drugs for more than 1 month, or blood pressure can be effectively controlled only after taking 4 or more antihypertensive drugs).
    9. Stroke, cerebrovascular accident or transient ischemic attack within 6 months prior to the first dose.
20. Pregnant or lactating women.
21. Any active serious mental illness, medical condition or other symptom/condition that, in the judgment of the investigator, may interfere with treatment, compliance or the ability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Up to 3 years.
  Assessing the incidence of adverse events (AEs) using the Common Terminology Criteria for Adverse Events (CTCAE Version 5)

SECONDARY OUTCOMES:
Assessment of the AUC of STI-8591 and its major metabolites (if any). | At the end of Cycle 1 and the first day of Cycle 2 (each cycle is 30 days) .
  Assessment of the pharmacokinetic profile of STI-8591 and its major metabolites (if any) in advanced AML:AUC(area under the concentration-time curve)
Assessment of the Tmax of STI-8591 and its major metabolites (if any). | At the end of Cycle 1 and the first day of Cycle 2 (each cycle is 30 days) .
  Assessment of the pharmacokinetic profile of STI-8591 and its major metabolites (if any) in advanced AML:Tmax (time to peak)
Assessment of the Cmax of STI-8591 and its major metabolites (if any). | At the end of Cycle 1 and the first day of Cycle 2 (each cycle is 30 days) .
  Assessment of the pharmacokinetic profile of STI-8591 and its major metabolites (if any) in advanced AML:Cmax(peak concentration)
Percentage change in FLT3 plasma inhibitory activity (PIA) relative to baseline | At the end of Cycle 1 and the first day of Cycle 2 (each cycle is 30 days) .
  Assessment of the percentage of biomarker changes relative to baseline for STI-8591 in advanced AML
Assessing the CRc of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:CRc, defined as CR, CRh and CRi as judged according to ELN2022 criteria.
Assessing the CR rate of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:CR rate, defined as the CR rate judged according to ELN 2022 criteria.
Assessing the objective remission rate ORR (CRc + PR + morphologic leukemia-free status [MLFS]) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:ORR, defined as CR, CRh, CRi, MLFS and PR as judged by ELN2022 criteria.
Assessing the duration of remission (DOR) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:DoR, defined as the time between the subject's first achievement of ORR and the first detection of recurrent disease, treatment failure, or death from any cause, whichever occurs first.
Assessing the event-free survival (EFS) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:EFS, defined as the time from the start of the subject's enrollment to the occurrence of any event (treatment failure/relapse after CR, CRh or CRi/permanent termination of treatment for any reason/death from any cause), whichever occurs first.
Assessing the progression-free survival (PFS) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:PFS, defined as the time between the subject's first study treatment and the onset of treatment failure or death from any cause, whichever occurs first.
Assessing the leukemia-free survival (LFS) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:LFS, defined as the time between the first attainment of CRc and the first detection of recurrent disease or death from any cause, whichever occurs first.
Assessing the overall survival (OS) of STI-8591 in advanced AML. | Through study completion, an average of 2 years.
  Assessing the initial effectiveness of STI-8591 in advanced AML:OS, defined as the time between the subject's first study treatment and death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang, China